CLINICAL TRIAL: NCT01655160
Title: Effects and Mechanisms of Treatment Intensity of Mirror Therapy in Patients With Subacute Stroke: Outcomes in Brain and Movement Reorganization, Sensorimotor and Daily Functions, and Measures of Physiological Markers.
Brief Title: Effects and Mechanisms of Treatment Intensity of Mirror Therapy in Patients With Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100-4548B
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke rehabilitation; Mirror therapy; Functional performance; Kinematic analysis; Functional magnetic resonance image; Motor recovery
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mirror therapy treatment (Experimental): Three groups will be involved in this part of the whole project:MT with low-intensity group (MT-LI), MT with moderate-intensity group (MT-MI), MT with high-intensity group (MT-HI)
  Interventions: Behavioral: MT with low-intensity group (MT-LI); Behavioral: MT with moderate-intensity group; Behavioral: Mirror therapy with high intensity group
- control intervention group (Active Comparator): The part of this project will involve 1 treatment groups:control intervention group (CI)
  Interventions: Behavioral: Control intervention group

INTERVENTIONS:
Behavioral: MT with low-intensity group (MT-LI) — The MT-LI group will receive a 30-minute MT per session followed by a 30-minute functional training.
  Other Names: MT-LI
  Arms: mirror therapy treatment
Behavioral: MT with moderate-intensity group — The MT-MI group will receive a 60-minute MT per session followed by a 30-minute functional training.
  Other Names: MT-MI
  Arms: mirror therapy treatment
Behavioral: Mirror therapy with high intensity group — The MT-HI group will receive a 90-minute MT per session followed by a 30-minute functional training
  Other Names: MT-HI
  Arms: mirror therapy treatment
Behavioral: Control intervention group — The CI group will carry out a 30-minute conventional stroke rehabilitation training per session followed by a 30-minute functional training.
  Other Names: CI
  Arms: control intervention group

SUMMARY:
The purpose of this study will evaluate the long-term benefits, optimal dose and mechanisms of mirror therapy and its effects on physiological markers.

DETAILED DESCRIPTION:
This trial is to examine whether (1) the immediate effects of treatment intensity in MT would occur on sensorimotor impairments and functional performance in patients with subacute stroke; (2) the long-term benefits of treatment intensity in MT on functionality can persist for six months after treatment finished; and (3) the MT could result in cortical/movement reorganization as well as the changes in physiological markers.

ELIGIBILITY:
Inclusion Criteria:

* first episode of stroke in cortical regions
* time since stroke less than 3 months
* initial motor part of UE of FMA score ranging from 24 to 52
* no serious cognitive impairment

Exclusion Criteria:

* aphasia
* visual impairments
* major health problems or poor physical conditions
* currently participation in any other

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline, change from baseline in FMA at 2 weeks, and change from baseline in FMA at 4 weeks
  The UE subscale of the FMA (max. score 66) uses a 3-point ordinal scale to assess motor impairment.
Action Research Arm Test (ARAT) | Baseline, change of ARAT at 2 weeks, and change of ARAT at 4 weeks
  ARAT will be used to assess the motor function of UE. A total of 19 items are to test the movement of grasp, grip, pinch, and gross motor, with a scale of 0-3 for each item (maximal of 57).
Motor Activity Log (MAL) | Baseline, change of MAL at 2 weeks, and change of MAL at 4 weeks
  The MAL is a semi-structured interview of patients to assess the amount of use (AOU) and quality of movement (QOM) of the affected upper extremity in 30 important daily activities using a 6-point ordinal scale. Higher scores indicate better performance.
ABILHAND Questionnaire | Baseline, change of ABILHAND Questionnaire at 2 weeks, and change of ABILHAND Questionnaire at 4 weeks
  ABILHAND questionnaire is an inventory of 56 manual activities that uses a 3-point ordinal scale to measure subjectively perceived difficulty in performing everyday bimanual activity.
Adelaide Activities Profile (AAP) | Baseline, change of AAP at 2 weeks, and change of AAP at 4 weeks
  AAP will be applied to indicate the level of participation in household and community activities. This profile includes 21 activities in the four areas: domestic chores, household maintenance, service to others, and social activities.

SECONDARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) | Baseline and change of fMRI at 4 weeks
  uses the blood oxygenation level-dependent (BOLD) response to evaluate the brain reorganization after intervention.
Physiological marker measures | Baseline and change from baseline in physiological marker measures at 4 weeks
  measure inflammatory markers, oxidative stress markers, and erythrocyte deformability.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Kwei-shan, Toayuan County, Taiwan